CLINICAL TRIAL: NCT00125060
Title: Transesophageal MRI in Conjunction With Lipid Lowering Measures
Brief Title: Transesophageal Magnetic Resonance Imaging (MRI) in Conjunction With Lipid Lowering Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Surgi-Vision Inc (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 03-12-17-04; M681-217-84250
Record Dates: First submitted 2005-07-28; First posted 2005-07-29 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Heart Diseases
Keywords: Aorta; Atherosclerosis; MRI; statin; inflammatory markers
MeSH Terms: conditions — Heart Diseases; Atherosclerosis | interventions — Simvastatin

INTERVENTIONS:
Drug: Simvastatin (20mg versus 80mg/day)

SUMMARY:
This research is being done to investigate the ability of an experimental imaging method - transesophageal magnetic resonance imaging (TEMRI), to detect the change in aortic atherosclerotic plaque burden and morphology between patients on high dose cholesterol lowering medications and patients on standard dose cholesterol lowering medications. This study will use TEMRI to see how atherosclerosis (cholesterol build up) changes with cholesterol lowering medications. This study will also investigate whether these cholesterol-lowering medications will change levels of blood tests, called inflammatory markers, in patients' blood. People with atherosclerosis may join this study. This study will also store blood samples for future studies of cardiac diseases; no gene testing will be done.

DETAILED DESCRIPTION:
Using a new MRI coil developed by Hopkins researchers, the investigators are now able to image aortic atherosclerotic plaques in exquisite detail. This coil is placed into the esophagus via a small nasogastric tube and positioned next to the descending thoracic aorta. Using this method of transesophageal MRI (TEMRI), the investigators are able not only to measure the extent of aortic atherosclerosis and the size of individual plaques, but they can now image in such detail as to obtain information about plaque composition. The extent of aortic atherosclerosis has been correlated with cardiovascular events including heart attack and stroke. The investigators now propose to use this new imaging technique to study the effect of aggressive lipid lowering measures on patients with aortic atherosclerosis.

They plan to randomize patients with documented vascular disease to high dose (simvastatin 80mg) versus low dose (simvastatin 20mg) cholesterol lowering medications. The investigators expect to show a decrease in the extent of atherosclerosis, a change in plaque morphology and composition, and perhaps a decrease in cardiovascular events in the aggressive care group of patients.

They also plan to measure serum markers of inflammation in these patients at baseline and after therapy. C-reactive protein is the most studied of the markers that are independently correlated with cardiovascular events. The investigators hope to show that TEMRI correlates higher levels of C-reactive protein with more baseline atherosclerosis, and that treatment with high dose statin therapy reduces levels of inflammatory markers.

Finally they plan to store plasma collected on these patients to save for future studies of cardiac markers, which could then be correlated with the effect of statin therapy and the reduction in aortic atherosclerosis as documented by TEMRI.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Required to have documented atherosclerosis in at least 1 vascular territory defined as: at least moderate (>3.9mm) aortic atherosclerosis seen on transesophageal echocardiography; or moderate coronary artery disease (>50% lesion) in at least 1 coronary artery seen at cardiac catheterization; or >50% carotid lesion seen on ultrasound; or clinically documented peripheral vascular disease.

Exclusion Criteria:

* Patients could be on any statin therapy at entry, but not on a dose equivalent to or greater than 80mg of simvastatin.
* Patients with pacemakers, automated implanted cardioverter defibrillators (AICD), aneurysm clips, abnormal nasopharyngeal anatomy, active peptic ulcer disease, severe dysphagia, elevated baseline liver transaminases and serum creatinine (greater than 2 times the normal), decompensated congestive heart failure or inability to give informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2000-08; Study Completion 2004-04

PRIMARY OUTCOMES:
change in aortic atherosclerotic plaque area and volume on transesophageal and surface MRI

SECONDARY OUTCOMES:
serum levels of inflammatory markers like C-reactive Protein (CRP), Interleukin (IL-6), Tumor Necrosis Factor alpha(TNF-α)
cardiovascular events and stroke during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Joao AC Lima, MD, MBA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins - School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Result] Steen H, Warren WP, Desai M, Gautam S, Lai S, Heath S, Stuber M, Lima JA. Combined transesophageal and surface MRI provides optimal imaging in aortic atherosclerosis. J Cardiovasc Magn Reson. 2004;6(4):909-16. doi: 10.1081/jcmr-200036202. PMID 15646894
- [Result] Lima JA, Desai MY, Steen H, Warren WP, Gautam S, Lai S. Statin-induced cholesterol lowering and plaque regression after 6 months of magnetic resonance imaging-monitored therapy. Circulation. 2004 Oct 19;110(16):2336-41. doi: 10.1161/01.CIR.0000145170.22652.51. Epub 2004 Oct 11. PMID 15477398
- [Derived] Gottlieb I, Agarwal S, Gautam S, Desai M, Steen H, Warren WP, Xavier SS, Lima JA. Aortic plaque regression as determined by magnetic resonance imaging with high-dose and low-dose statin therapy. J Cardiovasc Med (Hagerstown). 2008 Jul;9(7):700-6. doi: 10.2459/JCM.0b013e3282f447c3. PMID 18545070